CLINICAL TRIAL: NCT03335748
Title: Is the Cogmed Program Effective for Youths With ADHD Under Pharmacological Treatment?
Brief Title: the Cogmed Program for Youths With ADHD
Acronym: ADHDtraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Université de Montréal (Other); Université de Sherbrooke (Other); Paris West University Nanterre La Défense (Other)
Responsible Party: Principal Investigator, Dentz Amélie, Ph.d, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UQAM 10
Record Dates: First submitted 2017-10-30; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: ADHD; ADHD - Combined Type
Keywords: ADHD; Combined type; Cognitive training; Intervention; Youths
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants were randomized into an experimental group that received the Cogmed program and an active control group that received a low-intensity comparison version of the training
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind evaluation Participant and assessor are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active control group (Active Comparator): The program for the active control group is the same as for the experimental group, except that the degree of difficulty of the exercises remains low and invariable across trials, with three items needing to be recalled throughout.
  Interventions: Other: Cognitive training Cogmed program
- the Cogmed program (Experimental): 12 exercises proposed in the Cogmed program. Eight of these target visuospatial WM and four target verbal WM. Eight exercises are preprogrammed for each session, for a total of 90 trials (Pearsons, 2014). The degree of difficulty of the trials increases as a function of the participant's performance. For each trial, the participant receives feedback on their performance.
  Interventions: Other: Cognitive training Cogmed program

INTERVENTIONS:
Other: Cognitive training Cogmed program — Cognitive training Cogmed program

SUMMARY:
The primary objective of this study was to examine the effects of the Cogmed training program on working memory among youths 7 to 13 years old, while controlling presence and presentation of ADHD-related comorbidity. A secondary objective was to examine the generalization of effects to ADHD symptoms, non-verbal reasoning, attentional and executive functions, motor impulsivity, reading comprehension, and mathematical reasoning. Participants were under pharmacological treatment for ADHD combined type and a comorbidity. They were randomized into an experimental group that received the Cogmed program and an active control group that received a low-intensity comparison version of the training. They were evaluated at three time points: six weeks prior to intervention onset (T1), immediately prior to onset(T2), and one week following intervention completion (T3).

DETAILED DESCRIPTION:
Participants completed the Cogmed WM training program at home.Each training session lasted from 30 to 45 minutes and was supervised by a parent. For five consecutive weeks, participants had to complete at least five sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* (1) be 7 to 13 years old;(2) had to be diagnosed with ADHD combined type and present a comorbid learning disability, oppositional defiant disorder or Tourette syndrome;and (3) had to be medicated for ADHD,

Exclusion Criteria:

* Youths were excluded from the study if diagnosed with epilepsy, an internalizing disorder (anxiety or mood disorder), an autism-spectrum disorder or mental retardation.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-02-22 (Actual); Primary Completion 2014-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
working memory | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  cognitive tests

SECONDARY OUTCOMES:
ADHD symptoms | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  questionnaire Child ADHD symptoms were assessed with the Conners 3AI questionnaire (Conners, 2008). The parent version for youths 6 to 18 years old was used. Each item is rated on a Likert scale from 0 to 3 (0=never or rarely; 1=sometimes; 2=often; 3=very often). The instrument's test-retest reliability and internal consistency have been found to be satisfactory, r=.84-.93, α=.80-.93. Expected outcome-Interventions to decrease symptom of ADHD (higher values represent a worse outcome).
  T score Guideline 70+Very Elevated Score 65-69 Elevated Score 40-59 Average score 60-64 High average score < 40 Low score Same guidelines are used for subscales. Subscales for inattention and Hyperactivity/impulsivity are used. Symptoms indicated for each subscale are summed to get the total.
non-verbal reasoning | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  cognitive tests
Attentional functions | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  cognitive tests
Motor impulsivity | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  cognitive tests
reading comprehension | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  academic achievement test
Executive functionning | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4
  Questionnaire The Behavior Rating Inventory of Executive Function (BRIEF; Gioia, Isquith, Guy, & Kenworth, 2000) was used. The parent version of the instrument comprises 86 items rated on a Likert scale from 0 to 2 (0= never or rarely; 1=sometimes; 2= often). The questionnaire's psychometric properties have been found to be adequate, with both internal consistency,α = .72-.98, and test-retest reliability,r= .82, reaching satisfactory levels. The Working Memory scale was used to measure daily WM.The Global Executive Function scale was used to assess the child's daily executive function at home and school.
  Expected outcome-Interventions to decrease executive dysfunction (higher values represent a worse outcome).
  Range : 65-100 Elevated Score 50-65 Average score < 50-0 Low score Same guidelines are used for subscales. Symptoms indicated for each subscale are summed to get the total.
mathematical reasoning | Change is being assessed to compare the effects of the Cogmed training program and an active control group. 6 weeks prior to intervention (T1),immediately prior to intervention (T2), Just after intervention (3) and six months after follow-up (4)
  academic achievement test

CONTACTS AND LOCATIONS:
Overall Officials: Marie-claude Guay, Pr, Study Director — Université du Quebec at Montréal
Locations (1):
- Dentz Amélie, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chacko A, Bedard AC, Marks DJ, Feirsen N, Uderman JZ, Chimiklis A, Rajwan E, Cornwell M, Anderson L, Zwilling A, Ramon M. A randomized clinical trial of Cogmed Working Memory Training in school-age children with ADHD: a replication in a diverse sample using a control condition. J Child Psychol Psychiatry. 2014 Mar;55(3):247-55. doi: 10.1111/jcpp.12146. Epub 2013 Oct 7. PMID 24117656
- [Result] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731